CLINICAL TRIAL: NCT06611826
Title: A Prospective, Single-arm Phase II Clinical Study of GEP (Gemcitabine, Recombinant Human Endostatin, and Carrellizumab) Combined With High-low-dose Radiotherapy in Non-locally Treatable Recurrent Nasopharyngeal Carcinoma
Brief Title: GEP Combined With Radiotherapy in Non-locally Treatable Recurrent NPC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-766（IIT）
Record Dates: First submitted 2024-08-23; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Nasopharynx Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Gemcitabine; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEP (Experimental): Gemcitabine, recombinant human endostatin and carrilizumab combined with high-low dose radiotherapy
  Interventions: Drug: GEP (Gemcitabine, Recombinant Human Endostatin, and Carrellizumab) Combined With High-low-dose Radiotherapy

INTERVENTIONS:
Drug: GEP (Gemcitabine, Recombinant Human Endostatin, and Carrellizumab) Combined With High-low-dose Radiotherapy — The R-GEP regimen is as follows: Gemcitabine (G; 1.0 g/m2, d1, d8) in combination with recombinant human vascular endothelial growth factor (E; 150 mg, continuous intravenous infusion for 72 hours) and Carelizumab (P; 200 mg), administered every three weeks for a total of six cycles. During the 2nd-4th cycles, low-dose radiotherapy is administered to modulate the immune microenvironment (R: one course of radiotherapy per cycle: including booster fractions of 1 Gy*3 times for the recurrent lesions, once a day, for three cycles). Approximately three weeks after the completion of the sixth cycle of GEP regimen (or the last cycle), high-dose fractionated radiotherapy (5-8 Gy*5 times, once a day) is given to the recurrent lesions. Immune maintenance therapy continues until one year after treatment completion or disease progression.
  Other Names: recombinant human endostatin

SUMMARY:
This research aims to assess both effectiveness and safety of combining R-GEP regimen comprising gemcitabine, recombinant human endostatin, and cerexinib with low- and high-dose radiotherapy in managing unresectable recurrent nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Eligible patients will undergo screening before enrolling in this trial 。 The participants will receive R-GEP therapy according to specified dosing schedules over six cycles. Additionally administered low-dose radiotherapy during specific cycles serves to modulate immune microenvironment while high-dose fractionated radiotherapy follows completion of GEP therapy courses. Maintenance immunotherapy continues up until one year post-treatment conclusion or disease progression.Finally, the participants were evaluated accordingly。

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years;
2. ECOG performance status 0-2;
3. Pathological or clinical imaging diagnosis of recurrent nasopharyngeal carcinoma;
4. With imaging assessable lesions (assessed by RECIST 1.1 criteria);
5. Recurrent lesions are not eligible for curative local treatment (including but not limited to extensive invasion of recurrent lesions; recurrent lesions with obvious necrosis or ulceration, with bleeding risk; recurrent lesions extensively invading surrounding nerves/vessels or skin/muscle; obvious late radiation therapy complications after previous treatment: radiation-induced brain injury, posterior cranial nerve injury, dysphagia, severe myofibrosis; second or multiple courses of radiation therapy after recurrence or multiple recurrences);
6. The following requirements must be met for the function of major organs:

   Hematological parameters tolerable to treatment: white blood cells ≥3.0×10^9/L, neutrophils ≥1.5×10^9/L, hemoglobin ≥9 g/dL, platelets ≥90×10^9/L.

   Liver and kidney function: ALT, AST <1.5 times the upper limit of normal (ULN), total bilirubin <1.5×ULN, serum creatinine (Cr) ≤1.5×ULN; Echocardiographic assessment, left ventricular EF ≥50%;
7. The patient has signed an informed consent form and is willing and able to comply with the visit schedule, treatment plan, laboratory tests, and other research procedures.
8. Voluntarily enroll in this study, sign an informed consent form, have good compliance and willingness to cooperate with follow-up.

Exclusion Criteria:

1. Subjects who cannot accept or tolerate chemotherapy or radiotherapy for various reasons;
2. Subjects who can be cured by definitive radiotherapy or surgery;
3. Subjects who have undergone major surgical procedures within the past 4 weeks or have not fully recovered from such procedures;
4. Subjects who are currently participating in other drug clinical trials;
5. Serious cardiac disease or discomfort, including but not limited to the following conditions:

   * History of congestive heart failure or impaired systolic function (LVEF <50%);
   * Uncontrolled high-risk arrhythmias, such as atrial tachycardia, resting heart rate >100bpm, significant ventricular arrhythmias (such as ventricular tachycardia) or higher-level atrioventricular conduction block (i.e., Mobitz Ⅱ second-degree atrioventricular conduction block or third-degree atrioventricular conduction block);
   * Angina requiring anti-angina drug therapy;
   * Clinically significant valvular heart disease;
   * ECG showing a penetrating myocardial infarction;
   * Uncontrolled hypertension (systolic blood pressure >180mmHg and/or diastolic blood pressure >100mmHg);
6. Subjects who have a history of hypersensitivity to any component of the study drug;
7. Any other situation in which the investigator deems the subject unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
3 year OS rate | 3 year
  3 year OS rate

SECONDARY OUTCOMES:
ORR | 3year
  ORR
DCR | 3year
  DCR
3 year PFS rate | 3 year
  3 year PFS rate